CLINICAL TRIAL: NCT00512499
Title: Osteoporosis and Peripheral Fractures: Treatment and Investigation Multidisciplinary at the chUS
Brief Title: Strategies to Treat Osteoporosis Following a Fragility Fracture
Acronym: OPTIMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Procter and Gamble (Industry); Sanofi (Industry); Novartis (Industry); Amgen (Industry); Eli Lilly and Company (Industry); Servier (Industry); Warner Chilcott (Industry)
Responsible Party: Principal Investigator, Gilles Boire, MD, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 06-091
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Osteoporosis; Fractures
Keywords: Osteoporosis; Fragility fractures; Fracture clinics; Orthopedic surgeons
MeSH Terms: conditions — Osteoporosis; Fractures, Bone | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Placebo Comparator): CONTROL GROUP (first year only; maximum 300 patients): patients seen by CHUS orthopedists at the Hotel-Dieu site, where no nurse coordinator is available for inclusion. This is random but not randomized.
  Interventions: Behavioral: Control group
- Group 2 (Active Comparator): MINIMAL INTERVENTION GROUP: 1/2 of patients, randomly selected.
  INTERVENTION: A nurse coordinator will identify patients with fragility fractures and inform the patient about osteoporosis as the cause of the fracture, the benefit of treatment, and the options of treatment adapted to the individual patient. Written information will be sent to his/her family physician containing a presumed osteoporosis diagnosis, investigation to be performed, correct interpretation of any osteodensitometry results in the context of a fragility fracture, the options of treatment, and alternatives if the first prescriptions are not tolerated or stopped. Intervention
  Interventions: Behavioral: Minimal Intervention
- Group 3 (Experimental): INTENSIVE INTERVENTION GROUP: 1/2 of patients, randomly selected Multiple layers of intervention will be added: results of the basic blood investigation for osteoporosis will be transmitted to the family physician with a personal letter explaining the importance of seeing the patient rapidly and indicating the urgency of initiating a treatment and indicating detailed instructions of treatment. The patient will be called at 4, 8, 12,16 and 24 months to monitor drug adherence, correct inadequate intake, and try to improve adherence. If the patient is not taking an adequate treatment at 4, 8 or 12 months, a letter will be sent again to the family physician asking to treat the patient according to recommendations.
  Interventions: Behavioral: Intensive Intervention

INTERVENTIONS:
Behavioral: Control group — Informing patient that fracture probably of fragility origin and suggesting to consult primary care practitioner. After 8 months, if not treated, Intensive intervention will be offered
  Arms: Group 1
Behavioral: Minimal Intervention — Multiple layers of intervention will be added: results of the basic blood investigation for osteoporosis will be transmitted to the family physician with a personal letter explaining the importance of seeing the patient rapidly and indicating the urgency of initiating a treatment and indicating detailed instructions of treatment. The patient will be called at 4, 8, 12,16 and 24 months to monitor drug adherence, correct inadequate intake, and try to improve adherence. If the patient is not taking an adequate treatment at 4, 8 or 12 months, a letter will be sent again to the family physician asking to treat the patient according to recommendations.
  Arms: Group 2
Behavioral: Intensive Intervention — INTENSIVE INTERVENTION GROUP: 1/2 of patients, randomly selected results of the basic blood investigation for osteoporosis will be transmitted to the family physician with a personal letter explaining the importance of seeing the patient rapidly and indicating the urgency of initiating a treatment and indicating detailed instructions of treatment. The patient will be called at 4, 8, 12,16 and 24 months to monitor drug adherence, correct inadequate intake, and try to improve adherence. If the patient is not taking an adequate treatment at 4, 8 or 12 months, a letter will be sent again to the family physician asking to treat the patient according to recommendations.
  Sequential serum will be stored frozen in order to measure levels of blood markers of bone metabolism (at a later date)
  Arms: Group 3

SUMMARY:
Osteoporosis is a very frequent and easily treatable disease. Rates of treatment of affected patients is very low, as few high risk patients initiate treatment and only a minority of those pursue treatment for long enough time to prevent fractures. Patients presenting a fragility fracture after 50 years of age are at high risk of osteoporosis and may represent the ideal group of patients in which intervention aimed at improving initiation and persistence on treatment will be most effective.

Our first hypothesis is that the availability of a dedicated nurse practitioner to identify patients with fragility fractures among patients presenting at fracture clinics of orthopedic surgeons will increase markedly the rate of identification of osteoporosis.

Our second hypothesis is that giving to both the patient and its primary health practitioner (PHP) the patient's clinical, biological and radiological data along with individualized care suggestions will yield significantly better results than giving to the patient and its PHP generic information on osteoporosis risk, investigation and treatment.

DETAILED DESCRIPTION:
3- The OPTIMUS INTERVENTIONS

3.1. PROGRAM GOALS and OBJECTIVES

The OPTIMUS program is a health intervention whose aim is to increase the rate of long-term treatment of osteoporosis in patients with incident fragility fractures by addressing both initiation of treatment and persistence on treatment. Participation to the program will be voluntary.

Specifically, the goals of OPTIMUS are:

1. To increase the rate of initiation of treatment of osteoporosis following a fragility fracture in patients presenting to the CHUS. This rate is currently of about 30% in the Province of Quebec, according to the Recognizing Osteoporosis and its Consequences in Quebec (ROCQ) survey.

   We hope to demonstrate that a coordinated approach combining successful identification of patients with fragility fractures evaluated at the CHUS, quality information to the patients and to family physicians, rapid and appropriate management and initiation of treatment (see below) of these patients by general practitioners will lead to appropriate levels of treatment of osteoporosis after an episode of fracture. Our objective is to initiate treatment within 8 months after fracture in at least 50% of such patients who accept to participate with Minimal Intervention, 75% with Intensive Intervention, and 90% with Immediate treatment. The specifics of each Intervention are detailed below.
2. Improve long-term adherence to treatment of osteoporosis following initiation of treatment after a fragility fracture. The current rate of persistence is 30-50% at 1 year, most loss of persistence occurring during the first months.

Initiating treatment of osteoporosis is important. However, long-term adherence to treatment of osteoporosis is very poor, with most discontinuation or erratic intake of medication observed during the first few months. Our objective is to maintain observance (i.e. intake of at least 80% of the doses of drugs according to patient questionnaires and to delivery of drugs by pharmacists) at one year in at least 80% of the patients who have initiated treatment. To that end, we will also evaluate whether disclosure of the results of measurements of blood markers of bone metabolism will influence patient adherence to treatment over time. The correlation of these measurements with results of phone follow up interviews and drug delivery by pharmacists as indicators of adherence will also be determined.

Our objectives with the Intensive and Immediate treatment Interventions imply that 60% of patients with a fragility fracture would be treated for at least 16 months (i.e. 80% of the 75% of patients who have initiated a treatment will adhere long-term). After 16 months of treatment, the rate of loss of adherence is likely to be lower, but information is lacking on that subject. We will partially address this question by following patients up to 2 years. Longer rates of adherence need to be ascertained, but this represents an objective that is not part of the current proposal.

Why setting these objectives at 60% of long-term adherence to treatment?

Our objective to treat 60% of the patients may appear quite low. However, it is significantly higher than the appalling 20-30% rate of initiation of treatment currently seen in the province of Quebec and in Canada in general, combined with the 30-50% long-term adherence observed in practice (translating currently into 5-20% of patients taking appropriate long-term treatment for osteoporosis). If we are successful, the rate of treatment will be increased by 3 to 10 times.

On the contrary, our objective to treat 60% of the patients may appear unrealistic. To attain this goal, we have to include all health practitioners involved in patients' care (e.g., family physician, orthopedist, pharmacist, and the patients themselves), as well as testing additional safety nets to ensure adherence, including patients' recall by the nurse coordinator, estimating the impact of adding the results of serum markers of bone metabolism, and allowing problematic patients (i.e. patients with hip fracture, those without family physicians, those with complex medical situations, and those who do not adhere despite all other measures) the possibility to obtain a consultation with a bone specialist.

Effect on fracture rates If our objective to treat 60% of the patients is attained, it is likely to translate into a significant reduction of close to 50% of vertebral fractures (a decrease of 80-90% of the risk of recurrent vertebral fracture by bisphosphonates in 60% of the population) and of close to 30% of non-vertebral fractures, including the hip (reduction of 50% of the risk by bisphosphonate use in 60% of the population). These fractures are associated with morbidity (chronic pain, invalidity) and increased mortality, and contribute to increase the costs to the public Health Care System (hospitalization, surgery, rehabilitation, short-, mid- and long-term care in nursing homes needed). However, this impact on fractures will only become evaluable through access to Quebec's Health Insurance Agency (RAMQ) databases (through the regional Health Agency), by comparing the rate of new fracture for patients compliant to the intervention relative to the patients who will refuse to give their informed consent to be included into the intervention (estimated to 10-15% of the patients with fractures) and to the patients who will not be compliant (estimated to 40% of the patients who will give their consent to participate). In addition, this effect on fracture rates will only become significant after a longer period (3-5 years) of observation.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years of age
* Fragility fracture
* Consulting an orthopedic surgeon at the CHUS for treatment of the fracture

Exclusion Criteria:

* No Primary Care Practitioner
* Severe co-morbidity requiring specialized care
* Failure to consent

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Actual)
Dates: Start 2007-02; Primary Completion 2013-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients pursuing an effective osteoporosis treatment | At one year after the clinical fracture
  Patients with fragility fracture seeing an orthopedic surgeon for care of the fracture are included. Patients are then followed up by phone to assess new fragility fractures and initiation and persistence on osteoporosis treatments

SECONDARY OUTCOMES:
Rate of recurrent fragility fractures according to the site of the inclusion fracture | Up to 4 years after clinical fracture

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Boire, MD MSc, Principal Investigator — Université de Sherbrooke; François Cabana, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bissonnette L, April PM, Dumais R, Boire G, Roux S. Atypical fracture of the tibial diaphysis associated with bisphosphonate therapy: a case report. Bone. 2013 Oct;56(2):406-9. doi: 10.1016/j.bone.2013.07.012. Epub 2013 Jul 17. PMID 23871749
- [Background] Gaboury I, Corriveau H, Boire G, Cabana F, Beaulieu MC, Dagenais P, Gosselin S, Bogoch E, Rochette M, Filiatrault J, Laforest S, Jean S, Fansi A, Theriault D, Burnand B. Partnership for fragility bone fracture care provision and prevention program (P4Bones): study protocol for a secondary fracture prevention pragmatic controlled trial. Implement Sci. 2013 Jan 24;8:10. doi: 10.1186/1748-5908-8-10. PMID 23343392
- [Result] Roux S, Cabana F, Carrier N, Beaulieu M, April PM, Beaulieu MC, Boire G. The World Health Organization Fracture Risk Assessment Tool (FRAX) underestimates incident and recurrent fractures in consecutive patients with fragility fractures. J Clin Endocrinol Metab. 2014 Jul;99(7):2400-8. doi: 10.1210/jc.2013-4507. Epub 2014 Apr 29. PMID 24780062
- [Result] Roux S, Beaulieu M, Beaulieu MC, Cabana F, Boire G. Priming primary care physicians to treat osteoporosis after a fragility fracture: an integrated multidisciplinary approach. J Rheumatol. 2013 May;40(5):703-11. doi: 10.3899/jrheum.120908. Epub 2013 Mar 15. PMID 23504379
- [Result] Sale JE, Jain R, Akilan K, Senior K, Beaton D, Bogoch E, Boire G, Beaulieu MC, Lightfoot D, Funnell L. What Do We Know about Individuals Who Are Assessed as Being at Moderate Risk for Future Fracture in Canada? Health (Irvine Calif). 2015 May;7(5):514-520. doi: 10.4236/health.2015.75061. PMID 26523214
- [Derived] Roux S, Gaboury I, Gionet-Landry N, Garant MP, Beaulieu MC, Carrier N, Cabana F, Boire G. Using a sequential explanatory mixed method to evaluate the therapeutic window of opportunity for initiating osteoporosis treatment following fragility fractures. Osteoporos Int. 2018 Apr;29(4):961-971. doi: 10.1007/s00198-017-4374-8. Epub 2018 Feb 14. PMID 29445831